CLINICAL TRIAL: NCT00006438
Title: Rocker Sole Kinetics and Kinematics
Brief Title: How Shoes With Rocker Soles Affect Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-0118; R01HD031989 (NIH)
Record Dates: First submitted 2000-11-03; First posted 2000-11-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-03

CONDITIONS: Diabetic Feet
Keywords: Rocker sole; Plantar pressure; Diabetic feet; Insensate feet; gait analysis; Pedorthics; Gait abnormalities
MeSH Terms: conditions — Diabetic Foot; Mobility Limitation

INTERVENTIONS:
Device: Shoes with Rocker Soles

SUMMARY:
The purpose of this study is to compare how 3 special types of shoes with rocker-shaped soles help people with foot deformities to walk better. This study will use modern gait lab techniques to measure the forces on the bottom of the feet and to examine whether there is any effect higher on the leg from the rocker soles.

DETAILED DESCRIPTION:
The rocker sole is the most commonly prescribed external shoe modification. Use of rocker soles has been based on theoretical considerations and empirical observations with minimal scientific study and validation. With the passage of the therapeutic shoe bill (PL-100-203, section 4072) authorizing Medicare coverage of shoes and shoe modifications for diabetics, it is important to have objective data regarding the effect of rocker soles. This cross-over study will randomize 46 subjects (40 sensate and 6 insensate) to a combination of 3 rocker soles. Patients will be evaluated at baseline and after 20 minutes wearing each rocker sole shoe design to determine the effect of the type of rocker sole on plantar pressure and gait.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Insensate individuals

Exclusion Criteria:

* History or physical findings of any trunk, back or lower extremity orthopedic or neurologic abnormalities
* Inability to walk
* Inability to follow verbal directions

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 1997-01; Study Completion 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Wertsch, M.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin Gait Lab, Milwaukee, Wisconsin, United States

REFERENCES:
- See also: Medical College of Wisconsin website — http://www.mcw.edu
- See also: Click here for more information about the National Institute of Child Health and Human Development (NICHD). — http://www.nichd.nih.gov/